CLINICAL TRIAL: NCT03306368
Title: Youth Opioid Recovery Support: A Developmentally-specific Intervention for Home Delivery of Extended Release Naltrexone
Acronym: YORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Potomac Health Foundations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00144092
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Opioid-Related Disorders
Keywords: OUD; XR-NTX; assertive outreach; youth
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (TAU) (No Intervention): Participants receiving treatment as usual post-residential detox. TAU clinic-based treatment receiving standard clinic-based XR-NTX.
- Youth Opioid Recovery Support (YORS) (Experimental): Youth Opioid Recovery Support consists of the following component:
  Home delivery of XR-NTX, family framework, assertive continuing care incorporates outreach, home delivery of evidence based psychosocial treatment and case management in a model that specifically targets engagement and motivation in youth, contingency management.
  Interventions: Behavioral: Youth Opioid Recovery Support

INTERVENTIONS:
Behavioral: Youth Opioid Recovery Support — The components of the Youth Opioid Recovery Support intervention are:
  XR-NTX, home delivery of XR-NTX, the family framework approach engages and empowers families, assertive continuing care incorporates outreach, home delivery of XR-NTX, contingency management.
  Arms: Youth Opioid Recovery Support (YORS)

SUMMARY:
Opioid addiction among youth (including both adolescents and young adults) is a growing health problem with catastrophic consequences for young people and their families. The current opioid epidemic disproportionately affects youth. Furthermore, compared to adults, adolescents and young adults tend to have poorer engagement in and response to treatment than older adults. Relapse prevention medications are the clear standard of care for the treatment of opioid addiction in adults, but the evidence base for effectiveness including implementation is not well-established in youth, and concerns from the field emphasize poor adherence and retention. Further there is no consensus regarding models of care, psychosocial treatments and platforms for delivery of medications. Extended release naltrexone (XR-NTX) has proven effectiveness in adults and is a promising pharmacotherapy for youth, but the field needs further clarification of its optimal use and delivery in this target population, in the context of developmentally informed models of care. There is inadequate current capacity for specialty opioid specific treatment that integrates pharmacotherapy (relapse prevention medication) with psychosocial treatment in a context that is youth welcoming and family empowering.

DETAILED DESCRIPTION:
While retention in youth opioid treatment has generally been poor, assertive outreach has not been standard. There may be models from other populations with elements worth considering, such as Assertive Community Treatment (ACT) for severe and persistent mental illness or Assertive Continuing Care (ACC) for adolescents with cannabis use disorders. These are programs providing wrap-around services that include home-based services and medication administration visits, assertive outreach, intense case management, family engagement in order to address engagement barriers. ACC has considerable developmental validity, has been used widely and been scaled by SAMHSA in broad implementations for youth SUDs (other than OUD). ACT has become a broad standard of care for adults with chronic severe mental illness such as schizophrenia, who struggle with non-adherence and poor outcomes in conventional treatment. ACT also typically includes a medication home-delivery component. Most states have also developed standard public sector reimbursement models for ACT. But very little work has been done to adapt or adopt these models to the population of youth with opioid addiction.

Furthermore, limitations on adherence to XR-NTX under non-research conditions have been a barrier to optimal effectiveness. One study reported that among 62 adult patients completing inpatient detoxification who received an XR-NTX prior to discharge, 55% returned for a second injection and 16% received a third injection. In the LA County evaluation, only 17% of the 171 adults who received an XR-NTX injection received their third injection. The investigators' first case series of 16 youth receiving XR-NTX for opioid addiction, the average total number of outpatient doses received within 4 months of outpatient treatment was 1.5, corresponding to 38% of the potential 4 monthly doses, with 25% dropping out before receiving any outpatient doses. A naturalistic study published by the investigators, of young adult opioid treatment with either buprenorphine or XR-NTX and high intensity psychosocial treatment support included 13 cases treated with XR-NTX. This cohort had 40% retention at 6 months, no difference between the buprenorphine and XR-NTX groups, with an average number of 3.1 outpatient doses received within 6 months, corresponding to 52% of the potential 6 monthly doses. And while 54% received a 3rd outpatient dose, this was a low-volume program that selected highly motivated patients willing to accept the requirements and burdens of frequent attendance and intensive structure, and included only those who had initiated outpatient treatment following inpatient treatment.

To address these gaps discussed above, the investigators propose N=45 (~5 pilot intervention cases prior to randomization; see protocol) participants with OUD to be randomized to treatment as usual (TAU) or YORs intervention, which incorporates XR-NTX into a developmentally informed, multi-component model of care - Youth Opioid Recovery Support (YORS; see protocol for additional detail on the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Young adults age 18-26 with OUD who present for an index episode of residential/inpatient opioid detoxification and seek treatment with XR-NTX at Mountain Manor Treatment Center (MMTC).

Exclusion Criteria:

* Liver function tests (LFTs) > 5x upper limit of normal
* Psychiatric or medical instability (eg suicidailty, psychosis, Sickle Cell disease with frequent crises, etc) that would preclude participation in the trial
* Living situation (location greater than 60 miles from the center, homelessness) that would preclude participation in the trial

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Number of weeks retained in treatment | Treatment week 1 to 24 weeks
  # of weeks participant remains in treatment after discharge from inpatient care
Number of weeks negative for opioid use | Treatment week 1 to 24 weeks
  Number of weeks participant tests negative for opiates and reports no use of opiates.

SECONDARY OUTCOMES:
Number of patients who linked to after care | Treatment week 0 to treatment week 4
  Percent of patients who successfully link to after care from inpatient to outpatient will be calculated using total number of patients who linked over total number of patients referred.
Number of XR-NTX doses received | Treatment week 1 to 24 weeks
  Total number of XR-NTX doses received within 24 weeks
Number of weeks negative for substances other than opiates | Treatment week 1 to 24 weeks
  Number of weeks participant tests negative for substances other than opiates and reports no use of other illicit substances.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Fishman, MD, Principal Investigator — Mountain Manor Treatment Center; Marc Fishman, MD, Principal Investigator — Potomac Health Foundation
Locations (1):
- Mountain Manor Treatment Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vo HT, Robbins E, Westwood M, Lezama D, Fishman M. Relapse prevention medications in community treatment for young adults with opioid addiction. Subst Abus. 2016 Jul-Sep;37(3):392-397. doi: 10.1080/08897077.2016.1143435. Epub 2016 Jan 28. PMID 26820059
- [Background] Vo HT, Burgower R, Rozenberg I, Fishman M. Home-based delivery of XR-NTX in youth with opioid addiction. J Subst Abuse Treat. 2018 Feb;85:84-89. doi: 10.1016/j.jsat.2017.08.007. Epub 2017 Aug 31. PMID 28867062
- [Background] Fishman MJ, Winstanley EL, Curran E, Garrett S, Subramaniam G. Treatment of opioid dependence in adolescents and young adults with extended release naltrexone: preliminary case-series and feasibility. Addiction. 2010 Sep;105(9):1669-76. doi: 10.1111/j.1360-0443.2010.03015.x. Epub 2010 Jul 9. PMID 20626723
- [Background] Wenzel K, Fishman M. Mobile van delivery of extended-release buprenorphine and extended-release naltrexone for youth with OUD: An adaptation to the COVID-19 emergency. J Subst Abuse Treat. 2021 Jan;120:108149. doi: 10.1016/j.jsat.2020.108149. Epub 2020 Sep 24. PMID 33303086
- [Background] Wenzel K, Selby V, Wildberger J, Lavorato L, Thomas J, Fishman M. Choice of extended release medication for OUD in young adults (buprenorphine or naltrexone): A pilot enhancement of the Youth Opioid Recovery Support (YORS) intervention. J Subst Abuse Treat. 2021 Jun;125:108306. doi: 10.1016/j.jsat.2021.108306. Epub 2021 Jan 26. PMID 34016297
- [Result] Fishman M, Wenzel K, Vo H, Wildberger J, Burgower R. A pilot randomized controlled trial of assertive treatment including family involvement and home delivery of medication for young adults with opioid use disorder. Addiction. 2021 Mar;116(3):548-557. doi: 10.1111/add.15181. Epub 2020 Aug 4. PMID 32621368